CLINICAL TRIAL: NCT02164032
Title: The Role of IntraNasal Insulin in Regulating HepaTic Lipid COntent in HUMANS a Randomized, Controlled, Double Blinded Trial
Brief Title: The Role of IntraNasal Insulin in Regulating HepaTic Lipid COntent in HUMANS
Acronym: INTO_humans
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Dr. Michael Krebs, Prof. MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: INTO_humans; 2013-004463-32 (EudraCT Number)
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — insulin, neutral; Proton Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin dilution buffer (Placebo Comparator): During a subsequent 4-week treatment phase subjects will be randomly assigned to receive intranasal insulin (40 IE) Actrapid (100IE/mL); two 0.1 ml puffs per nostril) or placebo (insulin dilution buffer Novo Nordisk; two 0.1 ml puffs per nostril) four times a day (in total 160 IE Actrapid per day) before each main meal and before going to bed. 40 IE IN insulin enhances insulin concentration in the CSF without any changes in systemic insulin and glucose concentration, and no risk for hypoglycemia.
  Ectopic lipid content and heart function will be assessed weekly by non-invasive 1H magnetic resonance spectroscopy.
  Interventions: Drug: Insulin Dilution Buffer (Novo Nordisk); Other: 1H magnetic resonance spectroscopy
- Intranasal Insulin administration (Active Comparator): During a subsequent 4-week treatment phase subjects will be randomly assigned to receive intranasal insulin (40 IE) Actrapid (100IE/mL); two 0.1 ml puffs per nostril) or placebo (insulin dilution buffer Novo Nordisk; two 0.1 ml puffs per nostril) four times a day (in total 160 IE Actrapid per day) before each main meal and before going to bed. 40 IE IN insulin enhances insulin concentration in the CSF without any changes in systemic insulin and glucose concentration, and no risk for hypoglycemia.
  Ectopic lipid content and heart function will be assessed weekly by non-invasive 1H magnetic resonance spectroscopy.
  Interventions: Drug: Intranasal insulin administration; Other: 1H magnetic resonance spectroscopy

INTERVENTIONS:
Drug: Intranasal insulin administration — intranasal insulin (40 IE) Actrapid (100IE/mL); two 0.1 ml puffs per nostril) or placebo (insulin dilution buffer Novo Nordisk; two 0.1 ml puffs per nostril) four times a day (in total 160 IE Actrapid per day) before each main meal and before going to bed. 40 IE IN insulin enhances insulin concentration in the CSF without any changes in systemic insulin and glucose concentration, and no risk for hypoglycemia
  Other Names: insulin Actrapid
  Arms: Intranasal Insulin administration
Drug: Insulin Dilution Buffer (Novo Nordisk) — intranasal insulin (40 IE) Actrapid (100IE/mL); two 0.1 ml puffs per nostril) or placebo (insulin dilution buffer Novo Nordisk; two 0.1 ml puffs per nostril) four times a day (in total 160 IE Actrapid per day) before each main meal and before going to bed. 40 IE IN insulin enhances insulin concentration in the CSF without any changes in systemic insulin and glucose concentration, and no risk for hypoglycemia
  Other Names: vehicle
  Arms: Insulin dilution buffer
Other: 1H magnetic resonance spectroscopy — 1H MR spectroscopy and imaging will be performed on the on on the 3.0-T Tim Trio System (Siemens Erlangen Germany). MR Spectroscopy and imaging measurements will last no more than 90 minutes all together.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a common human liver pathology, closely associated with the obesity pandemic and insulin resistance. In the insulin resistant state the liver remains sensitive to pro-lipogenic signals of insulin, which further promote lipid accumulation. Secretion of very-low-density-lipoproteins (VLDL), the main carriers of triglycerides (TG) in the plasma, is the principal pathway for the liver to mobilize and dispose of lipids. Thus, hepatic TG export must not be too low in order to prevent steatosis. Our preliminary data from animal experiments suggest that enhanced brain insulin signaling promotes hepatic VLDL secretion, and reduces lipid accumulation in the liver. It remains to be tested whether other insulin sensitive tissues, such as the myocardium or the skeletal muscle, are also affected. In humans, neuropeptides, including insulin, can be delivered to the brain via an intranasal (IN) route of administration, without causing relevant systemic side effects.

Therefore, we hypothesize that by enhancing brain insulin signaling using chronic IN insulin administration hepatic TG export increases and prohibits lipid accumulation in the liver and other insulin sensitive tissues, such as the myocardium and the skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* BMI 22 - 27 kg/m2
* Age between 18 - 65 years
* Male sex

Exclusion Criteria:

* smoking
* regular medication
* metabolic or liver illnesses
* tendency towards claustrophobia
* Chronic sinusitis, diagnosed nasal polyposis, diagnosed severe septum deviation
* metal devices or other magnetic material in or on the subjects body which will be hazardous for NMR investigation [heart pacemaker, brain (aneurysm) clip, nerve stimulators, electrodes, ear implants, post coronary by-pass graft (epicardial pace wires), penile implants, colored contact lenses, patch to deliver medications through the skin, coiled spring intrauterine device, vascular filter for blood clots, orthodontic braces, shunt-spinal or ventricular, any metal implants (rods, joints, plates, pins, screws, nails, or clips), embolization coil, or any metal fragments or shrapnel in the body].

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Changes in total lipid content in the liver | one week before & at baseline & 1,2,3 and 4 weeks after intranasal insulin administration
  1H magnetic resonance spectroscopy

SECONDARY OUTCOMES:
Changes of hepatic Lipid composition | one week before & baseline & 1,2,3 and 4 weeks after intranasal insulin administration
  1H magnetic resonance spectroscopy
Changes of myocardial lipid content | baseline, 2 and 4 weeks after intranasal insulin administration
  1H magnetic resonance spectroscopy
Changes of myocardial lipid composition | baseline, 2 and 4 weeks after intranasal insulin administration
  1H magnetic resonance spectroscopy
Changes of skeletal muscle lipid content | baseline, 2 and 4 weeks after intranasal insulin administration
  1H magnetic resonance spectroscopy
Changes of lipid composition in skeletal muscle | baseline, 2 and 4 weeks after intranasal insulin administration
  1H magnetic resonance spectroscopy
changes in heart function | baseline, 2 and 4 weeks after intranasal insulin administration
  magnetic resonance imaging

OTHER OUTCOMES:
Changes of parameters of glucose and lipid metabolism | one week before & baseline & 1,2,3 and 4 weeks after initiation of intranasal insulin administration
  fasting Glucose, HbA1c, Cholesterol, LDL, HDL, TGs, non-HDL Cholesterol, FFAs
Lipid composition in plasma | one week before & at baseline & 1,2,3 and 4 weeks after intranasal insulin administration

CONTACTS AND LOCATIONS:
Overall Officials: Michael Krebs, MD, Prof., Principal Investigator — Medical University of Vienna, Währinger Gürtel 18-20, 1090 Vienna, Austria
Locations (1):
- Medical University Of Vienna, Department of Internal Medicine III, Vienna, Vienna, Austria